CLINICAL TRIAL: NCT06909357
Title: Creation of an Infrastructure to Support Delivery of mHealth Interventions for Cancer Patients Throughout Florida
Brief Title: Creation of an Infrastructure to Support Delivery of mHealth Interventions for Cancer Patients
Acronym: Project mFLi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Florida Biomedical Research Program - James & Esther King (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: MCC-23179
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Demonstration Project 1 (No Intervention): Screening and recruitment of cancer patients for connection to evidence-based smoking cessation treatment. The goal of the first demonstration project is to develop a feasible and effective method for screening cancer patients for smoking, determining treatment eligibility, and offering treatment.
- Demonstration Project 2 (Experimental): Pilot RCT of Quitline vs. Mobile-Delivered Smoking Cessation Intervention for Cancer Patients. The goal of this pilot feasibility study is two-fold: to evaluate the performance of the platform itself and to provide preliminary data for a future efficacy trial.
  Interventions: Other: Quitline Treatment (QT); Other: App-based Treatment (mHealth)
- Demonstration Project 3 (No Intervention): Utilizing machine learning to process data obtained from demonstration projects 1 and 2. In Demonstration Project 3, we will utilize all data collected in Demonstration Projects 1 and 2 to conduct machine and deep learning methods.

INTERVENTIONS:
Other: Quitline Treatment (QT) — Tobacco Free Florida Quitline. 10-week supply of Combination Nicotine Replacement Therapy (NRT).
  Arms: Demonstration Project 2
Other: App-based Treatment (mHealth) — Fully automated digitally-delivered smoking cessation intervention targeted to cancer patients. 10-week supply of Combination Nicotine Replacement Therapy (NRT).
  Arms: Demonstration Project 2

SUMMARY:
Despite the deleterious impact of smoking upon cancer treatment outcomes, smoking prevalence remains alarmingly high among cancer patients. Thus, reducing smoking by cancer patients is a public health priority, but treatments to date have demonstrated limited efficacy. Mobile health (mHealth) interventions have the potential to improve treatment efficacy while also greatly extending reach. The goal of this infrastructure proposal is to build a resource to facilitate the creation of mHealth tools that address the tobacco treatment needs of cancer patients. This resource, which will be available to researchers throughout Florida, would fill a critical gap in mHealth capacity.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* ≥100 lifetime cigarettes.
* English-speaking.
* Report smoking ≥ 1 cigarette in past 30 days.
* Working smartphone.

Exclusion Criteria:

* Failure to electronically confirm participation within 14 days of randomization via electronic link sent to participant's smartphone.
* Currently pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Screening | At Baseline
  Our screening process will be deemed feasible if: 1) ≥ 90% of patients complete the screener, 2) the proportion of patients identified as smokers meets or exceeds the historical self-reported proportions at each institution, 3) the program correctly identifies eligible participants and subsequently presents automated advice to quit, 4) it offers an opportunity to enroll in smoking cessation treatment, and 5) ≥ 30% of eligible patients enroll in treatment.
Usability: mHealth | Up to 6 Months
  Usability will be measured 2 ways: I) ≥ 80% will score ≥ 70 on the Systems Usability Scale (SUS), 10-item measure, (scores 0-100) assessing learnability and usability. II) ≥ 80% rate app as easy to use (dichotomous Y/N).
Acceptability/Satisfaction: mHealth | Up to 6 Months
  Acceptability/Satisfaction will be measured 4 ways: I) ≥ 80 will score mean ≥ 3.0 Client Satisfaction Questionnaire (CSQ), 8-item measure, (1-4 scale). II) ≥ 80% mostly or extremely satisfied with app. III) ≥ 80% would recommend this app to a friend to quit smoking (dichotomous Y/N). IV) ≥ 80% rate quality of intervention as good or excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Damon Vidrine, DrPH, Principal Investigator — Moffitt Cancer Center; Vani Simmons, PhD, Principal Investigator — Moffitt Cancer Center
Locations (3):
- United States (3):
  - University of Miami, Coral Gables, Florida
  - University of Florida, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida